CLINICAL TRIAL: NCT00084812
Title: An Open-Labeled, Non-Randomized Phase I Study of Safingol Administered With Cisplatin in Patients With Advanced Solid Tumors
Brief Title: Safingol and Cisplatin in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-002; MSKCC-04002
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; safingol

ARMS (1):
- Safingol and Cisplatin (Experimental): Patients receive safingol IV over 1 hour and cisplatin IV over 1 hour on day 1. Courses repeat every 21 days* in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients receive safingol on days 1 and 8 and cisplatin on day 8 for course 1 only; course 1 is 28 days in duration.
  Cohorts of 3-6 patients receive escalating doses of safingol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated at that dose level.
  Interventions: Drug: cisplatin; Drug: safingol

INTERVENTIONS:
Drug: cisplatin
Drug: safingol

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Safingol may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of safingol when given with cisplatin in treating patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of safingol when administered with cisplatin in patients with locally advanced or metastatic solid tumors.

Secondary

* Determine the toxic effects of this regimen in these patients.
* Determine the clinical pharmacokinetics of this regimen in these patients.
* Determine, preliminarily, the therapeutic activity of this regimen in these patients.
* Determine a safe dose (i.e., near the MTD) for phase II evaluation of this regimen in these patients.
* Determine, preliminarily, the role of ceramide and S1P, relative to response and apoptosis, in patients treated with this regimen.

OUTLINE: This is an open-label, non-randomized, dose-escalation study of safingol.

Patients receive safingol IV over 1 hour and cisplatin IV over 1 hour on day 1. Courses repeat every 21 days* in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receive safingol on days 1 and 8 and cisplatin on day 8 for course 1 only; course 1 is 28 days in duration.

Cohorts of 3-6 patients receive escalating doses of safingol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated at that dose level.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Locally advanced or metastatic disease
* Refractory to standard therapy OR not amenable to standard therapy
* No known CNS metastasis or CNS primary

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC count ≥ 3,500/mm^3
* Hemoglobin ≥ 9.5 g/dL
* Haptoglobin ≥ 30 mg/dL
* No concurrent hemolysis or history of non-drug-induced hemolysis (e.g., spherocytosis)

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL
* PT and PTT normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No cardiac arrhythmias
* No congestive heart failure
* No myocardial infarction within the past 6 months

Other

* Not pregnant
* Negative pregnancy test
* No nursing during and for at least 2 months after study participation
* Fertile patients must use effective contraception during and for at least 2 months after study participation
* HIV negative
* No mental incapacity that would preclude giving informed consent
* No moderate-to-severe high-frequency hearing loss
* No persistent severe (grade 2) drug-induced peripheral neuropathy
* No known allergy to cisplatin or any other platinum-containing compound
* No serious or uncontrolled infection
* No other medical condition or reason that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy

Chemotherapy

* Prior cisplatin allowed
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin)

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* Recovered from all prior therapy
* No concurrent vitamins, antioxidants, herbal preparations, or supplements

  * Concurrent single tablet multivitamin allowed
* No other concurrent investigational medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose as assessed by NCI toxicity scale during 3-4 weeks of treatment | 2 years

SECONDARY OUTCOMES:
Response as assessed by RECIST criteria during 3-6 weeks of treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Archie N. Tse, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Dickson MA, Carvajal RD, Merrill AH Jr, Gonen M, Cane LM, Schwartz GK. A phase I clinical trial of safingol in combination with cisplatin in advanced solid tumors. Clin Cancer Res. 2011 Apr 15;17(8):2484-92. doi: 10.1158/1078-0432.CCR-10-2323. Epub 2011 Jan 21. PMID 21257722